CLINICAL TRIAL: NCT05199337
Title: A Single Arm, Open-Label, Phase 1/2 Study of ZN-d5 for the Treatment of Relapsed or Refractory Light Chain (AL) Amyloidosis
Brief Title: Phase 1/2 Study of ZN-d5 for the Treatment of Relapsed or Refractory Light Chain (AL) Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: K-Group Alpha, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZN-d5-003
Record Dates: First submitted 2022-01-09; First posted 2022-01-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Amyloidosis; AL Amyloidosis
Keywords: Amyloidosis; AL Amyloidosis; RRAL; BCL2 Inhibitor; t(11;14); ZN-d5; Light Chain Amyloidosis; Light chain (AL) Amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive ZN-d5 orally (PO), once (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ZN-d5

INTERVENTIONS:
Drug: ZN-d5 — ZN-d5 will be administered orally
  Other Names: Study Drug

SUMMARY:
This is a single arm, Open-Label, Phase 1/2 Study of ZN-d5 for the Treatment of Relapsed or Refractory Light Chain (AL) Amyloidosis.

DETAILED DESCRIPTION:
A Single Arm, Open-Label, Phase 1/2 Study of ZN-d5 for the Treatment of Relapsed or Refractory Light Chain (AL) Amyloidosis. The first part of the study is phase 1 dose-escalation and the second part will be phase 2.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of AL amyloidosis based on histopathology, the presence of characteristic appearance on electron microscopy, or mass spectrometry typing of amyloid.
2. Prior AL amyloidosis treatment and has received at least one, but no more than three lines of prior therapy;
3. At least 3 months from hematopoietic stem cell transplantation or the shorter of 60 days or 5 half-lives for biologics, small molecules, or investigational drugs prior to starting treatment;
4. Measurable disease defined by serum differential free light chain;
5. Assessment of t(11,14) status by FISH;
6. Eastern Cooperative Oncology Group performance status ≤2 ;
7. History of organ involvement
8. Adequate bone marrow function prior to first administration of study drug;
9. Adequate organ function;

Key Exclusion Criteria:

1. Presence of non-AL amyloidosis, including wild-type or mutated ATTR amyloidosis;
2. Diagnosis of multiple myeloma according to the 2014 International Myeloma Working Group diagnostic criteria;
3. Mayo 2012 Stage IV disease;
4. Cardiac involvement exclusions apply to some subjects, including heart failure and cardiac arrhythmias.
5. Prior treatment with other BCL-2 inhibitors;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 18 Months
  Incidence and severity of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Dose limiting toxicities | 18 Months
  Incidence of Dose-limiting toxicities (DLTs) observed in DLT evaluable subjects

SECONDARY OUTCOMES:
PK Parameter: Finding max concentration (Cmax) of ZN-d5 | 48 months
  Determine the maximum observed concentration (Cmax) of ZN-d5 collected in the plasma from subjects at different dose levels.
PK Parameter: Finding time to maximum concentration (Tmax) of ZN-d5 | 48 months
  The duration (in hours) it takes for ZN-d5 to reach the maximum concentration (or Cmax) collected in the plasma from subjects at different dose levels.
PK Parameter: Finding half-life of ZN-d5 | 48 months
  The time takes for half the drug concentration of ZN-d5 to be eliminated (Half-life) from the plasma that was collected from subjects at different dose levels
PK Parameter: Finding the Area Under the Curve (AUC) of ZN-d5 | 48 months
  The total exposure of ZN-d5 over time (AUC) from the plasma collected by the subject at different dose levels.
Assess the hematologic response to ZN-d5 | 48 months
  The number of Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), No Response (NR), Progressive Disease (PD) using the AL Amyloidosis Hematologic Response Criteria.
Duration and time to hematologic response to ZN-d5 | 48 months
  The rate of, duration of, and time to CR, modified Complete Response (mCR), CR+VGPR, and mCR+VGPR

OTHER OUTCOMES:
To assess potential biomarker of ZN-d5 | 48 months
  The number of peripheral B-Cells from blood tests

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — K-Group Alpha subsidiary of Zentalis Pharmaceuticals
Locations (21):
- United States (5):
  - University of Southern California, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Tulane University, New Orleans, Louisiana
  - Washington University, St Louis, Missouri
  - Tennessee Oncology, Nashville, Tennessee
- Australia (4):
  - Blackwater (Westmead) Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Bank of Cyprus Hospital, Nicosia, Cyprus
- National and Kapodistrian University of Athens, Athens, Greece
- Israel (4):
  - Rambam Hospital, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (2):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
- Spain (4):
  - ICO Badalona-H.U. Germans Trias i Pujol, Barcelona, Badalona
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Clinic de Barcelona, Barcelona
  - Clinico de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke M, Nieto M. AL Amyloidosis: Current Treatment and Outcomes. Adv Hematol. 2025 Mar 3;2025:7280805. doi: 10.1155/ah/7280805. eCollection 2025. PMID 40226119